CLINICAL TRIAL: NCT00571493
Title: Phase I/II Study of VELCADE®-BEAM and Autologous Hematopoietic Stem Cell Transplantation for Relapsed Indolent Non-Hodgkin's Lymphoma, Transformed or Mantle Cell Lymphoma
Brief Title: VELCADE®-BEAM and Autologous Hematopoietic Stem Cell Transplantation for Non-Hodgkin's Lymphoma, or Mantle Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0438-05-FB; Protocol# X05184 (Other Grant/Funding Number: Millennium)
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Non-hodgkin's Lymphoma; Mantle Cell Lymphoma
Keywords: non-hodgkin's lymphoma; mantle cell lymphoma; BEAM; Velcade
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell | interventions — Bortezomib; Carmustine; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib Dose Escalation (Experimental): The phase I section of the study will follow a standard 3 + 3 design to determine the maximum tolerated dose (MTD) of bortezomib when added to a standard BEAM (BCNU (carmustine), etoposide, cytarabine, melphalan) conditioning regimen followed by autologous hematopoietic stem cell transplantation (ASCT).
  After the MTD is defined, additional patients will enroll in Phase II to obtain preliminary estimates of survival using the Phase I regimen.
  Interventions: Drug: Bortezomib; Drug: BEAM (carmustine (BCNU), etoposide, cytarabine, melphalan)

INTERVENTIONS:
Drug: Bortezomib — Patients will receive bortezomib in four dose cohorts ( .8. 1.0, 1.3, 1.5 mg/m²). Patients will receive bortezomib on days -11, -8, -5, and -2 before infusion of autologous stem cells.
  Other Names: Velcade
Drug: BEAM (carmustine (BCNU), etoposide, cytarabine, melphalan) — All study patients will receive BEAM per the standard institution protocol:
  BCNU (carmustine): 300 mg/m²on day -5 etoposide 100 mg/m² twice daily on days -5, -4, -3, and -2 cytarabine 100 mg/m² twice daily on days -5, -4, -3, -2 melphalan: 140 mg/m² on day -1 before infusion of autologous stem cells.
  Other Names: B - Carmustine (BCNU) E - Etoposide. A - Cytarabine (Ara-C, cytosine arabinoside) M - Melphalan

SUMMARY:
This is a Phase I/II trial designed to study the toxicity and Maximum Tolerated Dose (MTD) of bortezomib in combination with BEAM (carmustine (BCNU), etoposide, cytarabine, melphalan) and autologous hematopoietic stem cell transplantation (ASCT) and to obtain a preliminary estimate of the response rate to this combination.

DETAILED DESCRIPTION:
Primary Objective:The primary objective of the study is to evaluate the toxicity and determine the maximum tolerated dose (MTD) of bortezomib when added to a standard BEAM (carmustine (BCNU), etoposide, cytarabine, melphalan) conditioning regimen followed by autologous hematopoietic stem cell transplantation (ASCT).

Secondary Objective: The secondary objective of the study is to obtain a preliminary estimate of the overall response rate (ORR), progression free survival (PFS), and overall survival (OS) with this regimen.

Enrolled subjects will receive bortezomib in combination with BEAM (carmustine (BCNU), etoposide, cytarabine, melphalan) and autologous hematopoietic stem cell transplantation (AHSCT). Phase I treatment will administer bortezomib in four dose cohorts,in addition to the BEAM and ASCT. Three patients will be accrued in each dose cohort with enrollment starting at dose cohort. These subjects will be evaluated to establish the maximum tolerated dose of bortezomib in combination with BEAM autologous peripheral blood stem cell transplantation. Once established, the maximum tolerated dose will be utilized in treating an additional 20 subjects.

Follow-Up: Data collected will be utilized to obtain a preliminary estimate of the overall response rate, progressions free survival and overall survival using this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Persistent, relapsed or refractory indolent non-Hodgkin's lymphoma (Follicular grade I, II, or III), non-Hodgkin's lymphoma, composite lymphomas with ≥ 50% of tumor showing follicular histology, transformed follicular, lymphoplasmacytic, marginal zone lymphoma, small Lymphocytic Lymphoma (including T-cell subtypes), or mantle cell lymphoma that is relapsed, refractory, or in PR1 or CR1 (MCL only for CR1).
* Age >19 years.
* Signed written informed consent.
* Expected survival duration of > six months.
* Karnofsky Performance Status > 70.
* Eligible patients must have: Liver functions < 3x upper limits of normal (ULN) unless due to disease; ANC > 500 cells/mm3 and Platelet Count > 50 mm3.
* Patients > age 60 or with clinical signs of heart disease must have ejection fraction ≥ 45% LVEF.
* Patients with clinical signs of pulmonary insufficiency must have DLCO to be measured at > 50% of predicted value.
* Able to collect > 1.2 X 106/kg CD34+ cell for transplantation.
* No serious disease or condition that, in the opinion of the investigator, would compromise the patient's ability to participate in the study.
* Female patients must not be pregnant or lactating.
* Male and female patients of reproductive potential must follow accepted birth control measures.

Exclusion Criteria:

* Patients who are HIV seropositive
* Serum creatinine >2.5mg/dL or calculated creatinine clearance ≤ 50ml/min
* Total bilirubin >3 times upper limits of normal (unless due to Gilberts disease or malignancy), ALT and AST >4 times the upper limits of normal
* Active infection at the time of transplant
* Myocardial infarction within 6 months prior to enrollment or has New York Hospital Association (NYHA) Class III or IV heart failure uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-04-14 (Actual); Primary Completion 2014-11-01 (Actual); Study Completion 2014-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Vose, MD, Study Chair — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at an academic medical center in the United States.
Groups:
- Phase 1: Bortezomib-0.8 mg/m²: Bortezomib dose - 0.8 mg/m² will be added to standard BEAM (carmustine (BCNU), etoposide, cytarabine, melphalan) regimen followed by autologous hematopoietic stem cell transplantation (ASCT).
- Phase 1: Bortezomib-1.0 mg/m²: Bortezomib dose - 1.0 mg/m² will be added to standard BEAM (carmustine (BCNU), etoposide, cytarabine, melphalan) regimen followed by autologous hematopoietic stem cell transplantation (ASCT).
- Phase 1: Bortezomib-1.3 mg/m²: Bortezomib dose - 1.3 mg/m² will be added to standard BEAM (carmustine (BCNU), etoposide, cytarabine, melphalan) regimen followed by autologous hematopoietic stem cell transplantation (ASCT).
- Phase 1: Bortezomib-1.5 mg/m²: Bortezomib dose - 1.5 mg/m² will be added to standard BEAM (carmustine (BCNU), etoposide, cytarabine, melphalan) regimen followed by autologous hematopoietic stem cell transplantation (ASCT).
- Phase II: Bortezomib-1.5 mg/m²; Phase II: Bortezomib-1.3 mg/m²; Phase II:Bortezomib-1.0 mg/m²: Obtain a preliminary estimate of the overall response rate (ORR), progression free survival (PFS), and overall survival (OS) with maximum tolerated dose regimen.
Period: Overall Study
Arm/Group | Phase 1: Bortezomib-0.8 mg/m² | Phase 1: Bortezomib-1.0 mg/m² | Phase 1: Bortezomib-1.3 mg/m² | Phase 1: Bortezomib-1.5 mg/m² | Phase II: Bortezomib-1.5 mg/m² | Phase II: Bortezomib-1.3 mg/m² | Phase II:Bortezomib-1.0 mg/m²
Started | 3 | 4 | 3 | 3 | 11 | 12 | 6
Completed | 3 | 4 | 3 | 3 | 11 | 12 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I/II: In Phase 1 of the study, bortezomib was administered in 4 dose cohorts: 0.8 mg/m², 1.0 mg/m², 1.3 mg/m² and 1.5 mg/m². Bortezomib was given on days -11, -8, -5, and -2. All study patients received BEAM conditioning: carmustine (BCNU) 300 mg/m² on day -5, etoposide 100 mg/m² twice daily on days -5, -4, -3, and -2, cytarabine 100 mg/m² twice daily on days -5, -4, -3, and -2, and melphalan 140 mg/m² on day -1 before infusion of autologous stem cells. The objective of phase 1 was to determine the maximum tolerated dose (MTD) of bortezomib in this setting. The MTD was defined by observing any nonhematologic transplantation-related toxicity higher than grade 2 on the Bearman scale occurring between day -11 and engraftment. After the MTD was defined, patients were enrolled in Phase II to obtain a preliminary estimate of overall response rate (ORR), progression-free survival (PFS), and overall survival (OS) using this regimen.
Arm/Group | Phase I/II
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] | 58 [34 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Bortezomib
Description: The maximum tolerated dose (MTD) is defined to be the dose cohort below which 3 of 6 patients experience dose limiting toxicity (DLT), or the highest dose cohort of 1.5 mg/m², if 2 DLT were not observed at any dose cohort.
Time Frame: 14 months
Population: The MTD in Phase I was initially determined to be 1.5 mg/m2 but was later decreased to 1 mg/m2.
Measure: Number; unit: mg/m²
Groups:
- Phase I; Phase II: Maximum Tolerated Dose (MTD) of Bortezomib
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 13 | 29
mg/m² | 1.5 | 1.0

2. Secondary Outcome: Preliminary Estimate of Overall Response Rate (ORR)
Description: To obtain a preliminary estimate of overall response rate (ORR). The overall response rate is calculated as the number of patients who achieved complete response (CR) and partial response (PR) divided by the total number of evaluable patients.
Time Frame: 100 day post autologous hematopoietic stem cell transplantation (ASCT), one year post ASCT
Population: One hundred days after autologous hematopoietic stem cell transplantation (ASCT), 40 participants were evaluable for response.
  At year one post ASCT, 38 participants were evaluable for response. Participants evaluable for the secondary endpoints (Phase II) are those who complete the transplant procedure.
Measure: Number; unit: participants
Groups:
- Phase II: Overall Response Rate: To obtain a preliminary estimate of overall response rate (ORR). The overall response rate will be estimated as the number of participants who achieve a complete response (CR) or partial response (PR) divided by the number of evaluable participants.
Arm/Group | Phase II: Overall Response Rate
Number analyzed (Participants) | 40
participants
  Overall Response Rate (100 days after transplant) | 38
  Overall Response Rate (1 year after transplant): number analyzed (Participants) | 38
  Overall Response Rate (1 year after transplant) | 33

3. Secondary Outcome: Progression-free Survival (PFS), and Overall Survival (OS)
Description: To obtain a preliminary estimate of PFS and OS. Overall survival (OS) is defined as time from the first chemotherapy administered on the transplant trial until death from any cause. Progression free survival (PFS)is defined as time from therapy until relapse, progression, or death from any cause.
Time Frame: one year post autologous hematopoietic stem cell transplantation (ASCT) , 5 years post ASCT
Population: There were 38 evaluable patients at one year post autologous hematopoietic stem cell transplantation (ASCT).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase II: Progression Free Survival and Overall Survival: To obtain a preliminary estimate of progression free survival (PFS), and overall survival (OS)
Arm/Group | Phase II: Progression Free Survival and Overall Survival
Number analyzed (Participants) | 38
percentage of participants
  Progression Free Survival 1 year after transplant | 83 [68 to 92]
  Overall Survival 1 year after transplant | 91 [79 to 96]
  Progression Free Survival 5 years after transplant | 32 [15 to 51]
  Overall Survival 5 years after transplant | 67 [50 to 79]

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Phase I: Intervention: In Phase I of the study, bortezomib will be administered in 4 dose cohorts: .8 mg/m2 , 1.0 mg/m2, 1.3 mg/m2, and1.5 mg/m2. Three patients will be accrued in each dose cohort with enrollment starting at dose cohort 1 (.8 mg/m2). Bortezomib will be given on days -11,-8, -5, and -2. All study patients will receive BEAM conditioning per our standard institution protocol: carmustine (BCNU) 300 mg/m2 on day -5,etoposide 100 mg/m2 twice daily on days -5, -4, -3, and -2, cyatabine100 mg/m2 twice daily on days -5, -4, -3, and -2, and melphalan 140 mg/m2 on day -1 before infusion of autologous stem cells. The objective of phase I is to determine the maximum tolerated dose (MTD) of bortezomib in this setting. After the MTD is defined, another 20 patients will be enrolled in the Phase II portion of this protocol to obtain a preliminary estimate of the response rate.
- Phase II: Survival: Patients enrolled to obtain a preliminary estimate of ORR, Progression-free survival, and overall survival (OS) using this regimen.
Arm/Group | Phase I: Intervention | Phase II: Survival
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/29
Other Adverse Events (participants affected / at risk) | 13/13 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Intervention (N=13) | Phase II: Survival (N=29)
adynamic ileus (Gastrointestinal disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Intervention (N=13) | Phase II: Survival (N=29)
Neutropenic Fever (Blood and lymphatic system disorders) | 10 (11) | 19 (20)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 9 (10)
Peripheral Neuropathy (Nervous system disorders) | 0 (0) | 6 (6)
Vasovagal syncope/orthostatic hypotension (Nervous system disorders) | 1 (2) | 7 (8)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Ileus (Gastrointestinal disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No